CLINICAL TRIAL: NCT06903533
Title: The Effect of Puzzle Activity on Nursing Students' Willingness to Work With Older Adults and Gerontological Nursing Competence
Acronym: Puzzle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zühal Erdoğan, RN, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025 -397
Record Dates: First submitted 2025-03-28; First posted 2025-03-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Puzzle Activity
Keywords: Puzzle Activity, Nursing Students, Nursing

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Puzzle Activity Group (Experimental): The puzzles, which include questions related to basic knowledge and concepts of gerontological nursing competence, are required to be solved over a period of three weeks.
  Interventions: Other: Puzzle Activity
- Control group (No Intervention): After explaining the purpose and implementation of the study to the nursing students in the control group, the "Descriptive Information Form," the "Willingness to Work with Older People Scale," and the "Gerontological Nursing Competence Scale" will be administered. No intervention will be applied to the control group. At the end of the third week, the "Willingness to Work with Older People Scale" and the "Gerontological Nursing Competence Scale" will be re-administered.

INTERVENTIONS:
Other: Puzzle Activity — After assigning the students to the intervention and control groups, a puzzle activity will be conducted with the intervention group following a lecture. In preparing the puzzles, the researchers will use free online puzzle-making tools (e.g., https://crosswordlabs.com/). The puzzles will include questions related to basic knowledge and concepts concerning gerontological nursing competence. During the puzzle-solving process, the researcher will be present in the classroom and provide guidance to students when needed. After students complete the puzzles, the researcher will project the puzzle on the presentation screen and evaluate the answers through interactive discussion with the students. Upon completion of each puzzle, the researcher will collect the puzzles from the students to prevent contamination between the intervention and control groups. A post-test will be administered to students at the end of the puzzle activity.
  Arms: Puzzle Activity Group

SUMMARY:
The study will be conducted using a parallel-group randomized controlled experimental design to determine the effect of a puzzle activity on nursing students' willingness to work with older adults and their competence in gerontological nursing. The study population will consist of second-year students (N=243) enrolled in the Faculty of Nursing at a university. The sample of the study will include at least 86 nursing students, with 43 students in the puzzle group and 43 students in the control group. The research will be carried out between March 2025 and June 2025. In this study, data will be collected using the "Descriptive Information Form," the "Willingness to Work with Older People Scale," and the "Gerontological Nursing Competence Scale."

DETAILED DESCRIPTION:
The study will be conducted using a parallel-group randomized controlled experimental design to determine the effect of a puzzle activity on nursing students' willingness to work with older adults and their gerontological nursing competence. The study group will consist of second-year students (N=243) enrolled in the Faculty of Nursing at a university. The G*Power program was used to calculate the sample size. In the reference study (Kaynak, S., Ergün, S., & Karadaş, A. (2023). The effect of crossword puzzle activity used in distance education on nursing students' problem-solving and clinical decision-making skills: A comparative study. Nurse Education in Practice, 69, 103618), it was determined that at least 86 students (43+43) were needed, with α = 0.05, 80% power, and an effect size of 0.615.

After assigning the students to the intervention and control groups, a puzzle activity will be conducted with the intervention group following a lecture. In preparing the puzzles, the researchers will use free online puzzle-making tools (e.g., https://crosswordlabs.com/). The puzzles will include questions related to basic knowledge and concepts concerning gerontological nursing competence. During the puzzle-solving process, the researcher will be present in the classroom and provide guidance to students when needed. After students complete the puzzles, the researcher will project the puzzle on the presentation screen and evaluate the answers through interactive discussion with the students. Upon completion of each puzzle, the researcher will collect the puzzles from the students to prevent contamination between the intervention and control groups. A post-test will be administered to students at the end of the puzzle activity.

ELIGIBILITY:
Inclusion Criteria:

* • Being a second-year nursing student

  * Volunteering to participate in the study

Exclusion Criteria:

Not taking the Geriatric Health Nursing course

* Having difficulty in understanding and speaking Turkish
* Incomplete or incorrectly answered data collection tools
* Willingness to withdraw from the study voluntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Willingness to Work with Older People Scale | Baseline
  The scale was developed by Fadayevatan and colleagues (2018) to determine medical students' willingness to work with older adults. The Turkish validity and reliability of the scale were conducted by Akpınar Söylemez and colleagues (2022) with nursing and medical students The scale consists of 4 sub-dimensions and 20 items. The scale is a six-point Likert-type scale, where items are scored from 1 = strongly disagree to 6 = strongly agree. The minimum score that can be obtained from the scale is 20, and the maximum score is 120. Scores for each sub-dimension and a total score are calculated. Higher scores indicate a greater willingness to work with older adults
Willingness to Work with Older People Scale | At the end of the third week,
  The scale was developed by Fadayevatan and colleagues (2018) to determine medical students' willingness to work with older adults. The Turkish validity and reliability of the scale were conducted by Akpınar Söylemez and colleagues (2022) with nursing and medical students The scale consists of 4 sub-dimensions and 20 items. The scale is a six-point Likert-type scale, where items are scored from 1 = strongly disagree to 6 = strongly agree. The minimum score that can be obtained from the scale is 20, and the maximum score is 120. Scores for each sub-dimension and a total score are calculated. Higher scores indicate a greater willingness to work with older adults
Gerontological Nursing Competence Scale | Baseline
  The scale was developed by Tohmola et al. (2021) to measure nursing students' competencies in geriatric care. The Turkish validity and reliability study was conducted by Aslan et al. (2024). The scale consists of 53 items and 11 subdimensions. The scale is a 4-point Likert-type scale and is rated as follows:1 = Strongly Disagree, 2 = Partially Disagree, 3 = Partially Agree, 4 = Strongly Agree. The minimum score that can be obtained from the scale is 53, and the maximum score is 212. As the level of competence increases, the score obtained from the scale also increases
Gerontological Nursing Competence Scale | At the end of the third week,
  The scale was developed by Tohmola et al. (2021) to measure nursing students' competencies in geriatric care. The Turkish validity and reliability study was conducted by Aslan et al. (2024). The scale consists of 53 items and 11 subdimensions. The scale is a 4-point Likert-type scale and is rated as follows:1 = Strongly Disagree, 2 = Partially Disagree, 3 = Partially Agree, 4 = Strongly Agree. The minimum score that can be obtained from the scale is 53, and the maximum score is 212. As the level of competence increases, the score obtained from the scale also increases

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)